CLINICAL TRIAL: NCT04616079
Title: A Randomized, Double-Blind, Placebo-Controlled, Single Ascending Dose Study of the Safety, Tolerability and Pharmacokinetics of REGN6490 in Healthy Volunteers
Brief Title: Ascending Dose Study of the Safety and Tolerability of REGN6490 in Healthy Volunteers
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Sponsor decision
Sponsor: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: R6490-HV-1946; 2020-003261-19 (EudraCT Number)
Record Dates: First submitted 2020-10-29; First posted 2020-11-04 (Actual); Last update posted 2021-11-11 (Actual); Status verified 2021-11

CONDITIONS: Healthy Volunteer

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (8):
- IV Cohort 1 (Experimental): Single intravenous (IV) dose 1 of REGN6490 or matching placebo
  Interventions: Drug: REGN6490; Drug: Placebo
- IV Cohort 2 (Experimental): Single IV dose 2 of REGN6490 or matching placebo
  Interventions: Drug: REGN6490; Drug: Placebo
- IV Cohort 3 (Experimental): Single IV dose 3 of REGN6490 or matching placebo
  Interventions: Drug: REGN6490; Drug: Placebo
- IV Cohort 4 (Experimental): Single IV dose 4 of REGN6490 or matching placebo
  Interventions: Drug: REGN6490; Drug: Placebo
- IV Cohort 5 (Experimental): Single IV dose 5 of REGN6490 or matching placebo
  Interventions: Drug: REGN6490; Drug: Placebo
- SC Cohort 1 (Experimental): Single subcutaneous (SC) dose 1 of REGN6490 or matching placebo
  Interventions: Drug: REGN6490; Drug: Placebo
- SC Cohort 2 (Experimental): Single SC dose 2 of REGN6490 or matching placebo
  Interventions: Drug: REGN6490; Drug: Placebo
- SC Cohort 3 (Experimental): Single SC dose 2 of REGN6490 or matching placebo
  Interventions: Drug: REGN6490; Drug: Placebo

INTERVENTIONS:
Drug: REGN6490 — Single dose of REGN6490
Drug: Placebo — Placebo matching single dose of REGN6490

SUMMARY:
The primary objective of the study is to evaluate the safety and tolerability of single ascending intravenous (IV) and subcutaneous (SC) doses of REGN6490 in healthy adult participants

The secondary objectives of the study are to:

* Characterize the pharmacokinetic (PK) profile of single IV and SC doses of REGN6490 in healthy adult participants
* Assess immunogenicity of REGN6490 in healthy adult participants dosed with a single IV or SC dose of REGN6490

ELIGIBILITY:
Key Inclusion Criteria:

1. Body mass index between 18 and 31 kg/m2 (inclusive) at screening visit
2. Is judged by the investigator to be in good health based on medical history, physical examination, vital sign measurements, and ECG's performed at screening and/or prior to administration of initial dose of study drug
3. Is in good health based on laboratory safety testing obtained at the screening visit
4. Willing and able to comply with clinic visits and study-related procedures
5. Provide informed consent signed by study participant

Key Exclusion Criteria:

1. History of clinically significant cardiovascular, dermatological, respiratory, hepatic, renal, gastrointestinal, endocrine, hematological, psychiatric, or neurological disease, as assessed by the investigator, that may confound the results of the study or poses an additional risk to the participant by study participation
2. Presents any concern to the study investigator that might confound the results of the study or poses an additional risk to the participant by their participation in the study
3. Has any physical examination findings and/or history of any illness that, in the opinion of the study investigator, might confound the results of the study or poses an additional risk to the participant by study participation
4. Hospitalization (>24 hours) for any reason within 30 days of the screening visit
5. Is a current smoker, including e-cigarettes. Former smokers may be enrolled if they have stopped smoking for at least 3 months (90 days) prior to the screening visit

Note: Other protocol defined Inclusion/Exclusion criteria apply

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 57 (Actual)
Dates: Start 2020-11-19 (Actual); Primary Completion 2021-06-01 (Actual); Study Completion 2021-06-01 (Actual)

PRIMARY OUTCOMES:
Incidence and severity of Treatment-Emergent Adverse Events (TEAEs) | Up to Week 16
  TEAEs include abnormal laboratory testing, vital signs and electrocardiograms (ECGs)

SECONDARY OUTCOMES:
Serum Concentration of REGN6490 over time | Up to Week 16
Incidence of Treatment-Emergent REGN6490 Anti-Drug Antibodies (ADAs) | Up to Week 16

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trial Management, Study Director — Regeneron Pharmaceuticals
Locations (1):
- Regeneron Study Site, Ghent, Belgium

IPD SHARING:
Plan to Share IPD: Yes
All Individual Patient Data (IPD) that underlie publicly available results will be considered for sharing.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Individual anonymized participant data will be considered for sharing once the indication has been approved by a regulatory body, if there is legal authority to share the data and there is not a reasonable likelihood of participant re-identification.
Access Criteria: Qualified researchers may request access to anonymized patient level data or aggregate study data when Regeneron has received marketing authorization from major health authorities (eg, FDA, European Medicines Agency (EMA), Pharmaceuticals and Medical Devices Agency (PMDA), etc) for the product and indication, has the legal authority to share the data, and has made the study results publicly available (eg, scientific publication, scientific conference, clinical trial registry).
URL: https://vivli.org/